CLINICAL TRIAL: NCT02508779
Title: Blood Glucose Training for Women With Type 1 Diabetes Contemplating Pregnancy
Brief Title: BGAT (Blood Glucose Awareness Training) for Users Who Might Become Pregnant
Acronym: Bump2Be
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lee M Ritterband, Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17117; 5R21DK095206 (NIH)
Record Dates: First submitted 2015-07-21; First posted 2015-07-27 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 1; Pregnancy
Keywords: Diabetes; Blood Glucose Management; Preconception; Hypoglycemia; Women with diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bump2Be (Experimental): Blood Glucose Awareness Training for pregnancy or preconception
  Interventions: Behavioral: Bump2be
- Routine Care (Active Comparator): Routine care provided by subject's medical team
  Interventions: Other: Routine Care

INTERVENTIONS:
Behavioral: Bump2be — Bump2be is an internet intervention focusing on six topics (called cores) psycho-educational in nature with the goals of improving individuals' ability to: a) anticipate extreme BG levels, b) detect the presence of extreme BG levels, c) address current extreme BG levels, and d) prevent future extreme BG levels. The program includes didactic information, self-assessment tools, and active learning exercises.
  Arms: Bump2Be
Other: Routine Care — Participants will continue to receive care from their clinician.
  Arms: Routine Care

SUMMARY:
Ineffective management of blood glucose (BG) levels during preconception and pregnancy has been associated with severe maternal and fetal complications in women with type 1 diabetes (T1DM). Preconception care emphasizing stringent glycemic control in the preconception period and continued through early pregnancy can dramatically reduce these risks. However, the use of preconception care in the US has been disappointingly low due to a variety of organizational, provider, and patient centered factors. Furthermore, efforts to achieve tight glycemic control can increase the risk of severe hypoglycemia (SH) in T1DM women, potentially leading to serious health consequences. In this project, the investigators will test an education based Internet intervention (Bump2be or Blood glucose awareness training (BGAT) for users who might become pregnant) for use with T1DM women who are either actively trying to become pregnant (TP) or planning to become pregnant in the 12 months following their enrollment in this study (PP).

The main objective is to examine Bump2be's feasibility and preliminary efficacy as an intervention for these women to better regulate their BG levels and to meet their diabetes-related clinical targets for pregnancy. More specifically, Bump2be will be tested in a randomized clinical trial in which 58 T1DM women who are either TP or PP will be recruited. As part of this pre-post study design, participants will be randomly assigned to either the Bump2be intervention (n=29) or the routine care group (n=29). Data collected will include frequency of extreme BG, consequences of extreme BG, average BG levels (HbA1c level), estimation of BG, detection of low and high BG, and psychological functioning (including fear of hypoglycemia, avoidance of hyperglycemia, well-being, and internal locus of control). Interviews with up to 10 trial participants will be conducted at the conclusion of their study participation, to enable further optimization of the intervention in preparation for a subsequent R01 submission. This will be the first study investigating the use of the Internet to improve detection and management of extreme BG levels in Diabetes mellitus type 1 (T1DM) women who are either TP or PP.

DETAILED DESCRIPTION:
Scientific Background: The number of women with type 1 diabetes is expected to rise, particularly for those in their early reproductive years. Pre-existing diabetes in pregnancy can increase the risk of various maternal (e.g., hypoglycemia and diabetic ketoacidosis) and fetal complications. Uncontrolled BG levels immediately before and during pregnancy have been associated with miscarriage, pre-eclampsia, infant mortality and a twofold to fourfold increased risk of major congenital malformations. Maternal hyperglycemia has been shown to complicate pregnancy more than any other factor and has been associated with a higher rate of spontaneous abortions and congenital malformations. Preconception care emphasizing stringent BG control in the preconception period (at least three to six months prior to pregnancy) and continued throughout can significantly reduce these risks to levels that are similar to those reported for the non-diabetic population. These attempts to achieve tighter BG control have, however, been linked to increased incidence of SH in early pregnancy. These findings point to the critical importance of providing TIDM women with practical self-management skills that they can actively use to better manage their BG levels, and achieve their target glycemic control without undue risk of hypoglycemia in preparation for pregnancy. At present, however, there are no published behavioral interventions specifically tailored to improving detection and management of extreme BG levels in this patient population.

Rationale: The overall aim of this research is to develop (Phase 1) and test (Phase 2) the feasibility of the Bump2be Internet intervention for use with Diabetes mellitus type 1 (T1DM) women who are either TP or PP to help them effectively detect and reduce occurrences of extreme BG levels. Phase 1 of this research was submitted and approved by the Institutional Review Board (HSR# 16668) in 2013 and has been completed. The Bump2be intervention is based on BGATHome (Blood Glucose Awareness Training at Home), which is an automated, tailored, Internet delivered, psycho-educational intervention for T1DM patients. BGATHome is based on theories of self-regulation of health behavior, and the training focuses on patients' learning how to use both internal cues (e.g., physical and mood changes) and external cues (e.g., insulin and food action) to improve their BG awareness. It has proven successful in improving patients' glycemic control as well as their abilities to detect, anticipate, avoid, and treat extremes BG levels. Investigators have historically excluded T1DM women who were either pregnant or planning pregnancy from BGAT-related studies given their unique clinical needs and glycemic targets. The investigators now propose to evaluate the feasibility and effectiveness of Bump2be in women with T1DM who are either TP or PP to help them better regulate their BG levels and to meet the diabetes-related clinical targets for and during pregnancy. This protocol covers Phase 2 of this project.

Relevance: There is an urgent need to effectively support Diabetes mellitus type 1 (T1DM) women who are either TP or PP in their efforts to achieve and maintain strict glycemic control without experiencing SH. The investigators propose to test an Internet-based training program (Bump2be.org) to assist these women better anticipate, detect, manage, and prevent extreme BG occurrences to enable them to meet their glycemic goals for pregnancy. If found efficacious, Bump2be will be the first Internet-based behavioral intervention to train and assist these women achieve the recommended glycemic targets without increasing their risk of SH. The program has the potential to impact its target patients on a major public health level by supplementing their preconception care with a conveniently accessible program tailored to their specific needs. It holds promise to improve not only their BG management but also psychosocial functioning (e.g., reduced fear of hypoglycemia, improved diabetes-related quality of life and knowledge) with no additional burden on the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed with T1DM for at least a year
* Either actively trying to get pregnant or planning to become pregnant in the 12 months following enrollment in this study
* Own and routinely use a BG memory meter
* Measure BG more than twice per day
* Should be able to download personal BG meter onto a computer
* Be able to read and speak English
* Be able to provide informed consent
* Have regular access to a computer and the Internet, and be able to view the website content independently
* Reside in the United States

Exclusion Criteria:

* Residents of another country
* Unable to travel to Lab Corp for blood work

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-07; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Reduced frequency of extreme BG (as defined by the low and high BG index) | 3 months (during the intervention period)
Reduced consequences of extreme BG (e.g., diabetic ketoacidosis, SH) | 3 months (during the intervention period)

SECONDARY OUTCOMES:
Improved estimation of BG (as confirmed by BG Diary data) | 3 months (during the intervention period)
Improved detection of low and high BG (as confirmed by BG Diary data) | 3 months (during the intervention period)
Reduced fear of hypoglycemia (as confirmed by the Low Blood Sugar Survey) | Assessed pre and post intervention
Reduced extreme avoidance of hyperglycemia (as confirmed by the High Blood Sugar Survey) | Assessed pre and post intervention
Improved well-being (as confirmed by the Diabetes Distress Scale) | Assessed pre and post intervention
Improved internal locus of control (as confirmed by the Perceived Competence for Diabetes Scale and the Treatment Self-Regulation Questionnaire) | Assessed pre and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lee M Ritterband, PhD, Principal Investigator — University of Virginia Behavioral Health & Technology Laboratory
Locations (1):
- University of Viginia Center for Behavioral Health & Technology, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Cox D, Ritterband L, Magee J, Clarke W, Gonder-Frederick L. Blood glucose awareness training delivered over the internet. Diabetes Care. 2008 Aug;31(8):1527-8. doi: 10.2337/dc07-1956. Epub 2008 May 13. PMID 18477813
- [Background] Singh H, Owen S, Crook M, Gonder--Frederick L, Ingersoll & Ritterband L (2014) Women's experiences of pregnancy in type 1 diabetes: Implications for patient care. Annals of Behavioral Medicine, 47(Supplement 1): s17, A---054.
- [Background] Singh H, Murphy HR, Hendrieckx C, Ritterband L, Speight J. The challenges and future considerations regarding pregnancy-related outcomes in women with pre-existing diabetes. Curr Diab Rep. 2013 Dec;13(6):869-76. doi: 10.1007/s11892-013-0417-5. PMID 24013963